CLINICAL TRIAL: NCT04119869
Title: Feasibility and Acceptability of a Smart Phone Application Intervention to Enhance Coping for Young Adults With Cancer
Brief Title: Smart Phone App Intervention In Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Hanneke Poort PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-333
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Cancer; Young Adults; Behavioral Intervention; Smartphone Application
Keywords: Cancer; Young Adults; Behavioral Intervention; Smartphone Application
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iaya Smart Phone Application (Experimental): * Pre-study evaluation
  * Access to the smartphone intervention over the course of 12 weeks
  * Post-study evaluation and interview
  Interventions: Other: iaya

INTERVENTIONS:
Other: iaya — The iaya app is a smartphone application intervention that -through a variety of approaches, such as exercises aimed at identifying and changing thoughts and behaviors, imagery, and relaxation- seeks to enhance coping with the emotional impact of cancer.

SUMMARY:
This research study aims to explore the feasibility and acceptability of a smartphone application intervention, called iaya, among young adults with cancer.

DETAILED DESCRIPTION:
The iaya app was developed by clinicians from the Young Adult Program at the Dana-Farber Cancer Institute. The iaya app is a smartphone application intervention that -through a variety of approaches, such as exercises aimed at identifying and changing thoughts and behaviors, imagery, and relaxation- seeks to enhance coping with the emotional impact of cancer.

The investigators are conducting this study to see if the iaya app, specifically developed for young adults with cancer, is practical, to determine patient satisfaction with the iaya app, and to test study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-39 years
* Able to speak/read English
* Have a smart phone
* Receiving cancer treatment
* Active cancer care from an oncologist at Dana-Farber Cancer Institute

Exclusion Criteria:

* Neurological/cognitive condition interfering with the ability to understand and adhere to study procedures
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Number of participants who log in at least 10 times and open at least 3 coping skills exercises | 12 weeks
  Feasibility of iaya will be determined by calculating the percent of participants assigned to the iaya app who log in at least 10 times. Percent of participants assigned to the iaya app will open at least 3 coping skills exercises will also be considered as a component of feasibility.
Mean score on app usability questionnaire | 12 weeks
  Acceptability will be assessed with the 6-item app usability questionnaire rated on a Likert scale (0=strong disagree to 5=strongly agree). Items will prompt participants to rate the extend to which they would use this app frequently, found the app to be easy to use, well organized, learn how to use the app quickly, felt confident using the app, and if they found the app interactive. Scores can range from 0-30. Higher scores indicate higher perception of usability.

SECONDARY OUTCOMES:
Change in coping scores on the Cancer Behavior Inventory Brief Form | 12 weeks
  We will pilot the 12-item Cancer Behavior Inventory Brief Form (CBI-B) for future efficacy studies. The CBI-B measures self-efficacy for coping with cancer. Items are scored between 1 (not at all confident) to 9 (totally confident). Higher scores indicate a higher level of self-efficacy for coping with cancer.
  among young adults with cancer who had access to the iaya app for future efficacy studies.
Change in self-efficacy scores on the PROMIS Self-Efficacy for Managing Emotions Scale | 12 weeks
  We will pilot the 8-item PROMIS Self-Efficacy for Managing Emotions (PROMIS SEMEM) for future efficacy studies. The PROMIS SEMEM will be used to measure confidence to manage or control symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment, and anger. Items are scored on a scale from 1 (not at all confident) to 5 (very confident). Higher scores indicate a higher level of self-efficacy for managing emotions.
Change in emotional support on the PROMIS Emotional Support Scale | 12 weeks
  We will pilot the 12-item PROMIS Emotional Support (PROMIS ES) for future efficacy studies. The PROMIS ES measures perceived feelings of being cared for and valued as a person. Items are scores on a scale from 1 (never) to 5 (always). Higher scores indicate higher levels of perceived emotional support.
Change in quality of life on the Functional Assessment of Cancer Therapy-General Scale | 12 weeks
  We will pilot the 27-item Functional Assessment of Cancer Therapy-General (FACT-G) for future efficacy studies. The FACT-G consists of four sub scales: physical, emotional, social/family, and functional well-being. Items are scores between 0 (not at all) and 4 (very much). Higher scores indicate a higher level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Poort, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Hanneke_Poort@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

DOCUMENTS (1):
  • Informed Consent Form (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04119869/ICF_000.pdf